CLINICAL TRIAL: NCT00888329
Title: Prevention of Postoperative Nausea and Vomiting in a Gynecologic Surgery Population: A Randomized Placebo Controlled Trial of Aprepitant NK-1-receptor Antagonist
Brief Title: Aprepitant for Prevention of Postoperative Nausea and Vomiting in Elective Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Mayo Clinic (Other)
Responsible Party: Jennifer Klauschie MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-005478
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Elective hysterectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Experimental): 40 mg aprepitant
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — 40 mg administered orally with a sip of water prior to anesthesia induction.
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether 40 mg aprepitant administered before surgery is effective for preventing vomiting in the first 24 hours after surgery in women undergoing elective hysterectomy.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is the most frequent side effect after anesthesia, occurring in approximately 30% of unselected patients, and can be increased up to 70% in certain populations and procedures. Despite screening for patients at high risk for PONV, current prophylactic interventions fail to completely eliminate PONV for a substantial number of patients, leading to dehydration, electrolyte imbalance, prolonged hospitalizations, multiple doses of rescue therapy, and readmissions to the hospital (2). Aprepitant (Emend) is the first neurokin-1-receptor antagonist in a new class of antiemetics, which has already demonstrated powerful additive effects when combined with dexamethasone and a 5-HT3 to prevent both acute and delayed chemotherapy-induced nausea and vomiting (CINV). Early studies have also suggested it may useful in the prevention of postoperative nausea and vomiting (PONV).

Patients undergoing elective inpatient or outpatient hysterectomy will be offered enrollment in this prospective, randomized, double blinded, placebo controlled trial. Subjects will receive Aprepitant vs. placebo prior to induction of standardized anesthesia. Postoperative nausea (assessed with a VRS), vomiting, and use of rescue antiemetic therapy will be documented over a 48h period. Additionally, hospitalization days and readmissions for PONV will be compared. Adverse events will be reported to the IRB and manufacturer. By reducing PONV in a group of high risk patients, we anticipate a demonstrated decrease in rescue antiemetic costs and hospitalization days for PONV related issues.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective hysterectomy at Mayo Clinic in Arizona
* ASA I, II, or III

Exclusion Criteria:

* Pregnancy
* Concomitant bowel surgery other than appendectomy
* Hypersensitivity to study drug or rescue medication
* Preoperative score for nausea greater than 4 out of 10 points
* Severe hepatic insufficiency (Child-Pugh score > 9)
* Any condition which impairs the patient's ability to complete study assessments
* Intraoperative hemodynamic instability
* ICU admission
* Prolonged postoperative intubation
* Rifampin, carbamazepine, phenytoin, or other drugs which strongly induce CYP3A4 activity
* Other antiemetic within 12 hours prior to surgery
* Participation in a clinical trial using an investigational product

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Magrina, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began July 2007. Enrollment stopped October 2011 due to slow accrual.
Period: Overall Study
Arm/Group | Aprepitant | Placebo
Started | 125 | 131
Completed | 119 | 122
Not Completed | 6 | 9
Not completed — Physician Decision | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Placebo | Total
Number analyzed (Participants) | 50 | 70 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 53 (12) | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 70 | 120
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emesis
Description: This is the number of participants who had an episode of vomiting within 24 hours after emergence from anesthesia.
Time Frame: 24 hours after emergence from anesthesia
Population: ITT. However, the primary outcome measure was not recorded for 84 participants in the Aprepitant group and 63 participants in the Placebo group.
Measure: Number; unit: participants
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 35 | 59
participants | 6 | 17

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Aprepitant | Placebo
Serious Adverse Events (participants affected / at risk) | 3/34 | 2/37
Other Adverse Events (participants affected / at risk) | 15/34 | 20/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant (N=34) | Placebo (N=37)
anemia (Blood and lymphatic system disorders) | 1 | 0
blood clot in leg (Blood and lymphatic system disorders) | 1 | 0
hospital-aquired pneumonia (Infections and infestations) | 1 | 0
intestinal perforation (Injury, poisoning and procedural complications) | 0 | 1
wound infection (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant (N=34) | Placebo (N=37)
constipation (Gastrointestinal disorders) | 2 | 2
diarrhea (Gastrointestinal disorders) | 0 | 2
headache (Nervous system disorders) | 2 | 1
hot flashes (Endocrine disorders) | 2 | 1
nausea (Gastrointestinal disorders) | 2 | 1
paresthesia (Nervous system disorders) | 2 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 2
urinary tract infection (Infections and infestations) | 1 | 6
wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
wound infection (Infections and infestations) | 6 | 5

LIMITATIONS AND CAVEATS:
Results might have been influenced by selection bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes